CLINICAL TRIAL: NCT04679987
Title: Incidence of Paroxysmal Atrial Fibrillation (AF) in Patients With Acute Ischemic Stroke or Transient Ischemic Attacks (TIAs) by 48 Hours Holter Monitoring
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Badr Salem, Head of Critical care and emergency medicine, Helwan University
Other Study IDs: AFTIA
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Transient Ischemic Attack
Keywords: atrial fibrillation; transient ischemic attack
MeSH Terms: conditions — Ischemic Attack, Transient; Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- paroxysmal Af
  Interventions: Diagnostic Test: Holter ECG
- no paroxysmal Af
  Interventions: Diagnostic Test: Holter ECG

INTERVENTIONS:
Diagnostic Test: Holter ECG — all patients will be monitored for paroxysmal Af by holder ECG

SUMMARY:
200 patients presenting with symptoms of acute ischemic stroke or transient ischemic attack were included. All patients free of AF on presentation underwent 48 hours Holter monitoring within one week.

ELIGIBILITY:
Inclusion Criteria:

* patient with acute ischemic stroke or TIAs (within one week of onset)

Exclusion Criteria:

* history of persistent AF
* initial ECG is AF
* primary hemorrhagic stroke
* acute large vessel dissection
* inability or refusal of consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed as acute stroke or TIA in stroke unit and neurology outpatient clinic, neurology Department, faculty of medicine, Misr University for Science and Technology (MUST) University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
presence of paroxysmal Af | March 2019 -November 2020
  incidence of paroxysmal Af after TIA

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Badr, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No